CLINICAL TRIAL: NCT05443672
Title: A Multi-center Study of Breast Mass Screening and Diagnosis Using Deep Learning AI-based on Real-time Ultrasound Examination
Brief Title: Multi-center Study of Deep Learning AI in Breast Mass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Cancer Hospital & Institute (Other); Peking University Third Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Third Affiliated Hospital of Zhengzhou University (Other); Hebei Medical University Fourth Hospital (Other); Henan Cancer Hospital (Other Government); Shanxi Province Cancer Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Chongqing University Cancer Hospital (Other); Anqing Hospital affiliated to Anhui Medical University (Unknown); Qinhuangdao Maternal and Child Health Care Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Anyang Tumor Hospital (Other); The Third Affiliated Hospital of Jinzhou Medical University (Unknown); General Hospital of Jincheng Coal Industry Group (Unknown); Suzhou First People's Hospital (Unknown); Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: NCC2962
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Yizhun BUSMS — During the breast scanning, Yizhun BUSMS uses different color box to identify the breast lesion, and the box color indicates the risk grade of the lesion.

SUMMARY:
This multi-center study intends to evaluate the value of the detection and differential diagnosis of breast mass using deep learning AI-based real-time ultrasound examination.

DETAILED DESCRIPTION:
As the most common cancer expected to occur all over the world, extensive population screening plays a very important role in the early diagnosis and prognosis of the breast cancer. X-ray and ultrasound are the most commonly used screening methods, and ultrasound is especially important for Asian women with dense breasts. However, ultrasound is greatly affected by the operator's skill and experience, and the diagnostic accuracy varies greatly.

Artificial intelligence (AI) is a new method emerging in recent years, active in many medical fields and can effectively improve the diagnostic efficiency. However, previous researches on the application of AI in ultrasound are focused on single or multi-modality static ultrasound images. This multi-center study intends to evaluate the value of the detection and differential diagnosis of breast mass using deep learning AI-based real-time ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

1. Females who undergo ultrasound examination for a complaint of breast lesion;
2. The breast lesion that will obtain definite pathological diagnosis or follow-up at least two years.

Exclusion Criteria:

1. The breast lesion that has received CNB or FNA;
2. The breast cancer patient who has received neoadjuvant chemotherapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Femal patients with breast neoplasm
Sampling Method: Probability Sample
Enrollment: 1122 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of breast mass using deep learning AI-based real-time ultrasound examination | 12 months
  Pathology as a gold standard, to evaluate the diagnostic performance (sensitivity, specificity and accuracy)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Wang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No